CLINICAL TRIAL: NCT00045539
Title: A Phase II Study of Methotrexate and Thiotepa Chemotherapy for Patients With Newly Diagnosed Primary CNS Lymphoma
Brief Title: Methotrexate and Thiotepa in Treating Patients With Newly Diagnosed Primary CNS Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256605; NABTT-2109; JHOC-NABTT-2109
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-12

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Leucovorin; Methotrexate; Thiotepa

INTERVENTIONS:
Drug: leucovorin calcium
Drug: methotrexate
Drug: thiotepa

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate and thiotepa, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining methotrexate with thiotepa in treating patients who have newly-diagnosed primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete radiographic response in patients with newly diagnosed primary CNS lymphoma treated with methotrexate and thiotepa.
* Determine the duration of progression-free survival and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine whether tumor expression of BCL-6 is associated with response to this chemotherapy regimen and survival of these patients.
* Describe the relationship between initial response to steroids (if administered), response to this chemotherapy regimen, and survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive thiotepa IV over 15 minutes on day 1. Patients also receive methotrexate IV over 4 hours on days 1 (8 hours after thiotepa) and 14. Beginning 24 hours after the start of methotrexate infusion, patients receive leucovorin calcium IV or orally every 6 hours until rescue is achieved. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving disappearance of enhancement of disease on MRI receive an additional 28-day course followed by maintenance therapy comprising thiotepa and methotrexate once a month for 11 courses.

Patients undergo neuro-ophthalmologic exams annually for 2 years.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 23-39 patients will be accrued for this study within 8-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS lymphoma

  * Confirmed by 1 of the following:

    * Brain biopsy or resection
    * CSF cytology

      * Positive cytology or immunohistochemical diagnosis of monoclonality and measurable intracranial tumor
    * Vitreal biopsy
* Measurable and contrast-enhancing disease on the postoperative, pretreatment MRI or CT scan
* No radiographic evidence of ascites or pleural effusions

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* SGOT no greater than 4 times upper limit of normal

Renal

* Creatinine no greater than 2 mg/dL
* Creatinine clearance at least 50 mL/min

Other

* Mini mental score of at least 15
* HIV negative
* Able to achieve hydration
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ
* No allergy to methotrexate
* No serious infection
* No medical illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy or biologic therapy for this disease

Chemotherapy

* No prior chemotherapy for this disease
* No other concurrent chemotherapeutic agents

Endocrine therapy

* No prior hormonal therapy for this disease
* Prior glucocorticoid therapy allowed

Radiotherapy

* No prior radiotherapy for this disease
* No prior cranial irradiation

Surgery

* See Disease Characteristics

Other

* At least 1 week since prior salicylates, non-steroidal anti-inflammatory drugs, probenecid, folic acid, or sulfonamide medications
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Complete radiographic response

SECONDARY OUTCOMES:
Duration of progression-free survival and overall survival
Toxicity
Association of tumor BCL-6 expression with response
Relationship among initial response to steroids, response to chemotherapy, and survival

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, MPH, Study Chair — Massachusetts General Hospital
Locations (9):
- United States (9):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania